CLINICAL TRIAL: NCT06100718
Title: Discovery of New Cancer in the 1-year Follow-up After Ischemic Stroke in Patients at Risk: The INVISIBLE-1 Study
Acronym: INVISIBLE-1
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01797; 2021-01797 (Other: KEK-Number)
Record Dates: First submitted 2023-10-09; First posted 2023-10-25 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Cancer-related Stroke; Paraneoplastic Coagulopathy; Occult Cancer; Ischemic Stroke; Embolic Stroke of Undetermined Source; D-dimer
Keywords: Cancer-related stroke; D-dimer; ESUS; Occult cancer; Ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Acute ischemic stroke patients at high-risk for underlying occult cancer (elevated D-dimer and suspicion of ESUS at admission)

SUMMARY:
INVISIBLE-1 aims to prospectively follow patients up to one year after ischemic stroke to:

1. Determine the cumulative incidence of occult cancer in patients with embolic stroke of undetermined source (ESUS) and elevated D-dimer
2. Describe occult cancer characteristics and spontaneous course of occult cancer

Methodology

The investigators will include 370 stroke patients with elevated D-dimer (≥ 820 μg/L) at the time of stroke, suspicion of ESUS after initial workup and without known cancer. The investigators will perform a follow-up telephone interview at one year to assess the occurrence of a new cancer and characterize the course of the disease.

Significance

Determining the real incidence of occult cancer in high-risk patients will help support the implementation of screening trials in the future. Faster detection and treatment of occult cancers would significantly impact patient' outcomes by offering faster cancer treatment and optimal secondary stroke prevention.

DETAILED DESCRIPTION:
INVISIBLE-1 is the first prospective study conducting a 1-year post-stroke follow-up telephone interview in preselected stroke patients at high-risk for occult cancer.

INVISIBLE-1 aims to:

1. Prospectively determine the cumulative incidence of occult cancer in patients with elevated D-dimer and ESUS within 1 year after the ischemic stroke
2. Describe occult cancer characteristics and spontaneous course of occult cancer

Hypothesis

Elevated D-dimer and suspicion of ESUS at admission may predict an underlying unknown cancer at the time of index stroke. The investigators hypothesize that the cumulative incidence of newly diagnosed cancer within 1 year after stroke reaches 15% in patients presenting these characteristics. This percentage is higher than the 10% currently known according to available retrospective studies.

Project design

To ensure the recruitment of the majority of potential occult cancer patients, the investigators set the D-dimer cut-off for inclusion of ≥ 820 μg/L at admission, based on our intern retrospective analyses of 1001 patients (OCCULT-5 score). In patients with ESUS, this cut-off was associated with a sensitivity of 91% and a specificity of 56% for the presence of an occult cancer diagnosed within 1 year after the index-stroke.

As suggested by the current evidence, the investigators decided to set the limit for diagnosis of new cancer at 1 year after the index stroke. Beyond this period, the causality is questionable in our opinion.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature from patient or next of kin
* Age ≥ 18 years old
* Acute ischemic stroke with symptom onset within 48 h before admission
* Acute ischemic stroke with:

  * persistent signs and symptoms of stroke lasting for ≥ 24 hours OR
  * acute brain infarction documented by computer tomography (CT) or MRI
* D-dimer ≥ 820 μg/L measured after symptom-onset and within 24h after admission
* Embolic stroke of unknown source (ESUS)* after initial work-up (acute cerebral imaging, 12-lead electrocardiogram, cardiac monitoring for at least 24h and echocardiography)

Exclusion Criteria:

* Active cancer** known at time of index-stroke
* Intravenous Thrombolysis administrated prior to D-dimer measurement: Use of external laboratory value possible if available
* New diagnosis of central nervous system cancer
* Patient or next of kin (in case of lacking capacity) unlikely to be compliant or available for study follow-up interview

ESUS*: According to the definition from the NAVIGATE ESUS randomized trial: Non-lacunar ischemic stroke occurring in a patient in whom investigations did not show another specifically treatable underlying stroke etiology, primarily >50% stenosis in a proximal extracranial or intracranial artery, atrial fibrillation, other major-risk cardioembolic sources, or other determined etiology.

Active Cancer**: According to the definition from the International Society on Thrombosis and Haemostasis: Cancer diagnosed within the previous six months, recurrent, regionally advanced or metastatic cancer, cancer for which treatment had been administered within six months, or hematological malignancy that is not in complete remission for more than 5 years.

► Patients with history of cancer not meeting these criteria anymore can be included in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study aims to include 370 stroke-patients with elevated D-dimer (≥ 820 μg/L) at baseline and suspicion of ESUS after initial workup in emergency room.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with newly diagnosed cancer (occult cancer) | Within 1 year after ischemic stroke

SECONDARY OUTCOMES:
Determination of occult cancer characteristics | Within 1 year after ischemic stroke
  The description of the specific characteristics of occult cancers is defined by the location of the cancer, the histological type of cancer, the date of suspicion of cancer (e.g. via imaging), the type of investigation leading to the suspicion of cancer, the date of final diagnosis via histology, the presence of metastases at diagnosis, the type of treatment provided and the date of start of treatment.
Long-term functional outcome using the modified Rankin Scale (mRS) in stroke patients with occult cancer | At 1 year after ischemic stroke
  The mRS (ranging from 0-6) measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The higher the mRS score, the more disabled or dependent the patient (mRS 6 represents death).
All-cause mortality rate and cause-specific mortality rate | At 1 year after ischemic stroke
Rate of recurrent ischemic stroke, or systemic embolism in occult cancer-related stroke | Within 1 year after ischemic stroke
Stroke severity assessed with the National Institutes of Health Stroke Scale (NIHSS) score in patients with occult cancer | Baseline
  NIHSS score is used to quantify stroke severity. It ranges from 0 to a maximum of 42 points. The higher the score, the more extensive the stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Jung, MD, Principal Investigator — Inselspital, University of Bern
Locations (3):
- Switzerland (3):
  - Dept. of Neurology, Centre Hospital Universitaire Vaudois, Lausanne, Canton of Vaud
  - Dept. of Neurology, Universitätsspital Basel, Basel
  - Dept, of Neurology, Inselspital, University of Bern, Bern

IPD SHARING:
Plan to Share IPD: No